CLINICAL TRIAL: NCT04336384
Title: Impact of Covid-19 in Congenital Heart Disease - COVID-CHD
Brief Title: Impact of Covid-19 in Congenital Heart Disease
Acronym: COVID-CHD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Pr. Jean-Benoît THAMBO, Bordeaux (président) (Unknown); Dr. Céline GRUNENWALD GRONIER, Strasbourg (Unknown); Dr. Sébastien HASCOET, Le Plessis-Robinson (Unknown); Dr. Adeline BASQUIN, Rennes (Unknown); Dr. Nicolas COMBES, Toulouse (Unknown); Dr. Xavier IRIART, Bordeaux (Unknown); Dr. Daniela LAUX, Paris (Unknown); Dr. Magalie LADOUCEUR, Paris (Unknown); Pr. BERTRAND LEOBON, Toulouse (Unknown); Pr. Caroline OVAERT, Marseille (Unknown); Dr. Karine WARIN-FRESSE, Nantes (Unknown); Alexis BLANC, Montpellier (Unknown); Pr. Roland HENAINE, Lyon (Unknown); Hamouda ABASSI, Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0155
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-03

CONDITIONS: Congenital Heart Disease; Covid-19
Keywords: Congenital heart disease; Covid-19; Adults; Peadiarics
MeSH Terms: conditions — Heart Defects, Congenital; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ongoing Coronavirus (Covid-19) pandemic has recently generated the first epidemiological data on populations at risk. Currently, the risk factors, recognized for severe forms of Covid-19 infection, are elderly patients (> 70 years), obese patients, patients with chronic renal or respiratory diseases, cardiovascular history (stroke or coronary artery disease), high blood pressure, diabetes, and cancer.

The population of congenital heart disease (CHD) might also be at risk, however, no data is available in this group of patients.

CHD is the leading cause of birth defects, and as a result of recent medical advances, currently the number of adults with CHD exceeds the number of children, with an increasing prevalence of complex CHD. Approximately 200,000 children and 250,000 adults are living with a CHD in France today.

The French Society of Cardiology, coordinator of this study, issued recommendations on March 14, 2020 for the French CHD population on the basis of expert opinions based essentially on the data published in the general population. Nevertheless, there is a need to provide scientific data on the impact of Covid-19 in the pediatric and adult CHD population.

This study aims to assess the morbidity, the mortality and the risk factors associated with Covid-19 in patients with CHD in France

ELIGIBILITY:
Inclusion criteria:

* Patient with CHD as defined in the international classification ACC-CHD
* Covid-19 infection over the study period

Exclusion criteria:

- Patient with genetic heart disease (cardiomyopathy, hereditary rhythmic disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Peadiatric and adult patient with congenital heart disease and COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Covid-19 infection in the overall CHD population | through study completion, an average of 2 weeks
  Prevalence of Covid-19 infection in the overall CHD population

SECONDARY OUTCOMES:
Prevalence of Covid-19 infection per CHD sub-group | through study completion, an average of 2 weeks
  Prevalence of Covid-19 infection per CHD sub-group
Cardiovascular complications | through study completion, an average of 2 weeks
  Cardiovascular complications
Other complications | through study completion, an average of 2 weeks
  Other complications
Number of deaths | through study completion, an average of 2 weeks
  Number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD-PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Marelli AJ, Mackie AS, Ionescu-Ittu R, Rahme E, Pilote L. Congenital heart disease in the general population: changing prevalence and age distribution. Circulation. 2007 Jan 16;115(2):163-72. doi: 10.1161/CIRCULATIONAHA.106.627224. Epub 2007 Jan 8. PMID 17210844
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524